CLINICAL TRIAL: NCT03529942
Title: An Open-Label Study to Evaluate the Effect of the Administration of FX006 on Synovial Inflammation in Patients With Osteoarthritis of the Knee
Brief Title: Study to Evaluate the Effect of FX006 on Synovial Inflammation in Patients With OA of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX006-2017-014
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Pain; Intra-articular; Injection; Corticosteroid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — FX006; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FX006 32 mg (Experimental): Single intra-articular (IA) injection of FX006 32 mg
  Interventions: Drug: FX006 32 mg

INTERVENTIONS:
Drug: FX006 32 mg — Extended-release 32 mg FX006 IA injection
  Other Names: Zilretta

SUMMARY:
This is an open-label study assessing the effect of the administration of a single intra-articular (IA) injection of FX006 32 mg on synovial volume in patients with osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
This is an open-label study assessing the effect of the administration of a single intra-articular (IA) injection of FX006 32 mg on synovial volume in patients with osteoarthritis (OA) of the knee. The study will be conducted in male and female patients who are ≥ 40 years of age.

Eligible patients who provide written consent and meet all entry criteria will undergo initial ultrasound examination and MRI with contrast of the index knee, and then receive a single IA injection of FX006 administered to the index knee at Baseline/Day 1. Patients will return to the clinic at Weeks 6 and 24 for an MRI with contrast of the index knee and other assessments. Patients must also have a blood sample drawn for Estimated Glomerular Filtration Rate (eGFR) testing within 30 days prior to the scheduled MRIs. In addition, a patient questionnaire will be administered and adverse events (AEs) and concomitant medication updates will be collected via telephone at Weeks 12 and 18.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Male or female ≥ 40 years of age
* Body mass index (BMI) ≤ 40 kg/m^2
* Ambulatory and in good general health
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions
* Willing to abstain from use of protocol-restricted medications during the study
* Symptoms associated with OA of the index knee for ≥ 6 months prior to Screening (patient self-report is acceptable)
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA
* Kellgren-Lawrence (K-L) Grade 2 or 3 in the index knee based on X-ray performed during Screening (centrally read)

Exclusion Criteria:

* Any inflammatory arthritis including reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, gout or secondary OA from gout
* History of infection or crystal disease in the index knee joint
* Unstable index knee joint (such as a torn anterior cruciate ligament) within 12 months of Screening
* Surgery or arthroscopy of the index knee within 12 months of Screening
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA treatment of the index knee with hyaluronic acid (investigational or marketed) within 6 months of Screening
* IV or IM corticosteroids (investigational or marketed) within 3 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Any other IA drug/biologic in the index knee within 6 months of Screening or 5 half-lives (whichever is longer) (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy and amniotic fluid injection)
* Prior administration of FX006
* eGFR results <40 mL/minute
* Any contraindication to MRI Scanning (e.g., presence of certain ferromagnetic foreign bodies or electronic devices including most cardiac pacemakers, claustrophobia)
* Known hypersensitivity to any form of radiographic contrast
* Females who are pregnant or nursing or plan to become pregnant during the study; men who plan to conceive during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Study Director — Flexion Therapeutics
Locations (10):
- United States (9):
  - TriWest Research Associates, LLC, El Cajon, California
  - Biosolutions Research, La Mesa, California
  - Dream Team Clinical Research (formerly located in Anaheim), Pomona, California
  - Dream Team Clinical Research, Pomona, California
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - PMG Research, Inc. d/b/a PMG Research of Knoxville, Knoxville, Tennessee
- University of Leeds, Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- FX006 32mg: All patients who received any amount of FX006 32mg
Period: Overall Study
Arm/Group | FX006 32mg
Started | 129
Reached Week 6 With Paired MRI | 108
Completed | 106
Not Completed | 23
Not completed — Withdrawal by Subject | 13
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 7
Not completed — Needle inserted but no drug administered | 1
Not completed — Personal reasons | 1

BASELINE CHARACTERISTICS:
Population: All patients who received any amount of FX006 32mg
Groups:
- Total Population: All patients who received any amount of FX006 32mg
Arm/Group | Total Population
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 16
  White | 108
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 129

OUTCOME MEASURES:

1. Primary Outcome: Mean Standardized Change in Synovial Volume (SV) at 6 Weeks
Description: Synovial volume (mm^3) as measured by MRI and read by a central imaging vendor. Standardization was performed by dividing the model-derived least squares means and corresponding confidence intervals by the adjusted standard deviation (SD). Therefore, the mean standardized change represents the change in synovial volume expressed in standard deviation units.
Time Frame: Baseline to Week 6
Population: Participants with pre-treatment synovial volume measurement as determined by quantitative image analysis, as well as a quality Week 6 MRI who received a single intra-articular (IA) injection of FX006 32 mg
Measure: Least Squares Mean (95% Confidence Interval); unit: Standardized Units
Groups:
- Total Population: All patients who received a single intra-articular (IA) injection of FX006 32mg and had a pre-treatment synovial volume measurement
- Patients With Baseline Synovitis: The subset of the Total Population who had a pre-treatment synovial volume measurement of greater than 3000 mm^3 of gadolinium enhancement as determined by quantitative image analysis
Arm/Group | Total Population | Patients With Baseline Synovitis
Number analyzed (Participants) | 108 | 84
Standardized Units | -0.67 [-0.8131 to -0.5296] | -0.9 [-1.0573 to -0.7341]

2. Secondary Outcome: Mean Absolute Change in Synovial Volume at 6 Weeks
Description: Mean absolute change from baseline at 6 weeks in synovial volume (mm^3) as measured by MRI and read by a central imaging vendor. The least squares mean changes are estimated using a mixed effects model for repeated measures with fixed effects for study time point, study site, baseline score and baseline femur bone volume (mm^3) and a random effect for patient.
Time Frame: Baseline to Week 6
Population: Participants with pre treatment synovial volume measurement as determined by quantitative image analysis, as well as a quality Week 6 MRI who received a single intra-articular (IA) injection of FX006 32 mg
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Total Population | Patients With Baseline Synovitis
Number analyzed (Participants) | 108 | 84
mm^3 | -5469.68 (581.9123) | -7549.55 (683.6488)

3. Secondary Outcome: Mean Standardized Change in Synovial Volume (SV) at 24 Weeks
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: Participants with pre treatment synovial volume measurement as determined by quantitative image analysis, as well as a quality Week 24 MRI who received a single intra-articular (IA) injection of FX006 32 mg
Measure: Least Squares Mean (95% Confidence Interval); unit: Standardized Units
Groups:
- Total Population: All patients who received a single intra-articular (IA) injection of FX006 32 mg and had a pre-treatment synovial volume measurement
Arm/Group | Total Population | Patients With Baseline Synovitis
Number analyzed (Participants) | 88 | 68
Standardized Units | 0.20 [0.0536 to 0.3371] | 0.20 [0.0385 to 0.3618]

4. Secondary Outcome: Mean Absolute Change in Synovial Volume at 24 Weeks
Description: Mean absolute change (mm^3) from baseline at 24 weeks in synovial volume (mm^3) as measured by MRI and read by a central imaging vendor. The least squares mean changes are estimated using a mixed effects model for repeated measures with fixed effects for study time point, study site, baseline score and baseline femur bone volume (mm^3) and a random effect for patient.
Time Frame: Baseline to Week 24
Population: Participants with pre-treatment synovial volume measurement as determined by quantitative image analysis, as well as a quality Week 24 MRI who received a single intra-articular (IA) injection of FX006 32 mg.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Total Population | Patients With Baseline Synovitis
Number analyzed (Participants) | 88 | 68
mm^3 | 3239.94 (1184.5800) | 3476.52 (1408.7997)

ADVERSE EVENTS:
Time Frame: Through study completion; up to 28 weeks
Groups:
- Total Population: All patients who received an attempted single intra-articular (IA) injection of FX006 32 mg
Arm/Group | Total Population | Patients With Baseline Synovitis
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/129 | 1/102
Other Adverse Events (participants affected / at risk) | 31/129 | 28/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Population (N=129) | Patients With Baseline Synovitis (N=102)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Population (N=129) | Patients With Baseline Synovitis (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Thyroid Cyst (Endocrine disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Acute Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural Anxiety (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Synovial Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Cardiac Murmur (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
One patient experienced procedural anxiety during the placement of the syringe on the inserted needle and did not receive the full dose of FX006. This patient is still counted in the safety population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03529942/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT03529942/SAP_002.pdf
  • Informed Consent Form (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03529942/ICF_001.pdf